CLINICAL TRIAL: NCT00464230
Title: The Management of Intracapsular Fractures of the Proximal Femur. A Prospective, Randomized Trial of Two Parallel Screws and Hemiarthroplasty
Brief Title: Hemiarthroplasty or Internal Fixation for Displaced Femoral Neck Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-2005-OS
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2007-04

CONDITIONS: Femoral Neck Fractures
Keywords: Displaced Femoral Neck Fractures; Treatment; Function; Pain; Quality of life; Complications; Reoperations; Internal Fixation; Hemiarthroplasty; Activities of Daily Living
MeSH Terms: conditions — Femoral Neck Fractures; Pain | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Bipolar hemiarthroplasty (Charnley/Hastings)
Procedure: Internal fixation with two parallel screws (Olmed)

SUMMARY:
An estimated 1.6 million patients sustain a hip fracture every year, about half of these are intracapsular femoral neck fractures. A femoral neck fracture is a life changing event for any patient, and the risk of disability, increased dependence and death is substantial. The main treatment options for displaced femoral neck fractures are internal fixation and arthroplasty. It is established that there are more complications and reoperations after internal fixation, but there is no consensus about which procedure that gives best functional results.

DETAILED DESCRIPTION:
We plan to include patients with displaced intracapsular femoral neck fractures. The patients will be randomized by means of closed numbered envelopes to operation groups:

1. Two parallel screws (Olmed).
2. Hemiarthroplasty with Charnley/ Hastings prosthesis. A priori one would expect that there would be less morbidity and mortality with the less extensive and quicker operation with parallel screw and that a faster and better rehabilitation would be achieved with hemiarthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Displaced femoral neck fracture
* Age 60 or above
* Able to walk (any aids allowed)

Exclusion Criteria:

* Anesthesiologically unfit for arthroplasty surgery
* Previous symptomatic hip pathology (i.e. arthritis)
* Pathological fracture
* Delay of more than 96 hours from injury to treatment
* Not living in hospital area

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2002-09; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score at 4, 12 and 24 months
Barthel ADL Index at 4, 12 and 24 months
Eq-5d (Euroqol) at 4, 12 and 24 months

SECONDARY OUTCOMES:
Mortality
Re-operations
Complications
Morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Jan Erik Madsen, MD, PhD, Study Chair — Orthopedic Center, Ulleval University Hospital
Locations (1):
- Orthopedic Center, Ulleval University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Waaler Bjornelv GM, Frihagen F, Madsen JE, Nordsletten L, Aas E. Hemiarthroplasty compared to internal fixation with percutaneous cannulated screws as treatment of displaced femoral neck fractures in the elderly: cost-utility analysis performed alongside a randomized, controlled trial. Osteoporos Int. 2012 Jun;23(6):1711-9. doi: 10.1007/s00198-011-1772-1. Epub 2011 Oct 14. PMID 21997224
- [Derived] Frihagen F, Nordsletten L, Madsen JE. Hemiarthroplasty or internal fixation for intracapsular displaced femoral neck fractures: randomised controlled trial. BMJ. 2007 Dec 15;335(7632):1251-4. doi: 10.1136/bmj.39399.456551.25. Epub 2007 Dec 4. PMID 18056740